CLINICAL TRIAL: NCT01990248
Title: ZeSS: A Prospective Observational Safety Study of Patients With BRAF-V600 Mutation-positive Unresectable or Metastatic Melanoma Treated With Vemurafenib (Zelboraf®)
Brief Title: An Observational Safety Study in Zelboraf (Vemurafenib)-Treated Patients With BRAF-V600 Mutation-Positive Unresectable or Metastatic Melanoma (ZeSS)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: GP28492
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, prospective, observational safety study will evaluate the safety and effectiveness of Zelboraf (vemurafenib) in a real world setting. Data from Zelboraf-treated patients with BRAF-V600 mutation-positive unresectable or metastatic melanoma will be collected for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of the age of 18 years or older
* Diagnosis of BRAF-V600 mutation-positive unresectable or metastatic melanoma confirmed by a validated test and being treated with vemurafenib
* Vemurafenib treatment must have been initiated at the time of enrollment or no more than one month prior to enrollment
* Patient (or legally acceptable representative) has personally signed and dated the informed consent document indicating that he or she has been informed of all pertinent aspects of the study, if applicable
* Patient is willing to provide information on at least one alternate contact person for study staff to contact regarding the patient's whereabouts, should the patient become lost to follow-up during the course of the study

Exclusion Criteria:

* Patient was treated with vemurafenib as part of a clinical trial or expanded access program
* Patient has participated in any studies involving any investigational study drug within one month prior to initiating vemurafenib treatment
* Patient has any significant history of disease of medical condition (except metastatic melanoma) which in the judgment of the investigator has the potential to impact participation on the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable or metastatic melanoma treated with vemurafenib
Sampling Method: Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2013-03-23 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-07-26 (Actual)

PRIMARY OUTCOMES:
Incidence of non-cutaneous squamous cell carcinoma | 2 years
Incidence of cutaneous squamous cell carcinoma | 2 years
Incidence of QT prolongation (defined as QTc >500 ms or an increase in QTc >60 ms) | 2 years
Incidence of abnormal liver function | 2 years

SECONDARY OUTCOMES:
Incidence of a second (or subsequent) primary melanoma | 2 years
Incidence of gastrointestinal polyps | 2 years
Incidence of adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (80):
- Austria (3):
  - LKH Feldkirch; Onkologie, Feldkirch
  - Ordensklinikum Linz Elisabethinen ; Dermatologie, Linz
  - Krankenhaus Hietzing Wien, Vienna
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - CHIREC Edith Cavell, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
- Czechia (3):
  - FN Ostrava; Dermatology dep, Ostrava
  - University Hospital Prague, Prague
  - Komplexni onkologicke centrum Krajske nemocnice T. Bati, a.s. Zlin, Zlín
- Germany (31):
  - Klinikum Augsburg; Hauttumorzentrum, Augsburg
  - Charite- universitatsmedizin Berlin; Med. Klinik mit Schwerpunkt Hamatologie und Onkologie, Berlin
  - Ruhr-Universität Bochum; Klinik für Dermatologie und Allergologie, Bochum
  - Universitatsklinikum Bonn; Klinisches Studienzentrum Klinik fur Dermatologie, Bonn
  - Medizinisches Zentrum, Bonn
  - Dermatologisches Zentrum am Elbe Klinikum Buxtehude, Buxtehude
  - DRK Krankenhaus Chemnitz-Rabenstein; Hautkrebszentrum Chemnitz, Chemnitz
  - Universitätsklinikum "Carl Gustav Carus"; Klinik und Poliklinik fur Dermatologie, Dresden
  - Universitätsklinikum Düsseldorf; Hautklinik, Düsseldorf
  - Dermatologie und Allergologie HELIOS Hauttumorzentrum Erfurt, Erfurt
  - Universitatsklinikum Essen; Klinik für Dermatologie, Essen
  - SRH Wald-Klinikum Gera; Zentrum fur klinische Studien (ZKS), Gera
  - Universitaetsmedizin Goettingen; Abteilung Dermato-Onkologie, Göttingen
  - Universitätsmedizin Greifswald; Klinik und Poliklinik für Hautkrankheiten, Greifswald
  - Univ.- Hautklinik Heidelberg, Heidelberg
  - Friedrich-Schiller-Universitaet Jena; Klinik fuer Dermatologie und dermatologische Allergologie, Jena
  - Klinikum Kassel GmbH; Hauttumorzentrum HTZ, Kassel
  - Studienzentrum UnterEms; Onkologische Schwerpunktpraxis Leer; Dr. med. Lothar Müller, Leer
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH; Hauttumorzentrum Rheinpfalz, Ludwigshafen
  - UKSH Universitatsklinikum Schleswig-Holstein; Studienzentrum Dermatologie 10d, Lübeck
  - Klinik und Poliklinik fur Dermatologie; Universitatsklinikum Mainz, Mainz
  - Med. Fakultat Mannheim der Universitat Heidelberg; Klinik fur Dermatologie, Mannheim
  - Johannes Wesling Klinikum Minden;Haut Tumor Centrum Minden, Minden
  - Universitätsklinikum Münster; Klinik für Hautkrankheiten; Allgemeine Dermatologie und Venerologie, Münster
  - Fachklinik Hornheide; Abteilung für Dermatologie, Münster
  - Klinikum Nürnberg Nord; Hautklinik; Klinik für Dermatologie, Nuremberg
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Standort Quedlinburg; Hautkrebszentrum Harz, Quedlinburg
  - Klinikum Vest; Behandlungszentrum Kanppschaftskrankenhaus Recklinghausen, Recklinghausen
  - Universitätsmedizin Rostock; Klinik und Poliklinik für Dermatologie und Venerologie, Rostock
  - Eberhard-Karls-Universitat Tubingen; Sektion Dermatologische Onkologie, Tübingen
  - Universitätsklinikum Würzburg; Klinik und Poliklinik für Dermatologie Venerologie u. Allergologie, Würzburg
- Galway University Hospital; Clinical Trials Department, Galway, Ireland
- Italy (13):
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Policlinico S. Orsola Malpighi;Dip. Ematologia, Oncologia e Medicina di Laboratorio, Bologna, Emilia-Romagna
  - Ausl Ravenna-Osp.Infermi; Day Hospital Oncologia Medica, Faenza, Emilia-Romagna
  - Universita di Modena e Reggio Emilia;Dipartimento di Oncologia ed Ematologia, Modena, Emilia-Romagna
  - Ospedale "Guglielmo da Saliceto";U.O. Medicina Oncologica, Piacenza, Emilia-Romagna
  - Azienda ASL di Rimini (Presidi di Rimini - Cattolica)) - Ospedale degli Infermi;U.O. Oncologia, Rimini, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Oncologia, Pavia, Lombardy
  - A.O.V.V. - P.O. di Sondrio; S.O.C. Oncologia Medica, Sondrio, Lombardy
  - A.U Careggi di Firenze;Oncologia, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliera Universitaria Senese, U.O.C. Immunoterapia Oncologica, Siena, Tuscany
- Netherlands (4):
  - Amphia Ziekenhuis, locatie Langendijk;Oncology, Breda
  - Academ Ziekenhuis Groningen; Medical Oncology, Groningen
  - Atrium MC, Parkstad Heerlen; Poli Interne, Heerlen
  - Maastricht University Medical Center,Division of Medical Oncology; Dept. Internal Medicine, Maastricht
- Poland (6):
  - Centrum Onkologii w Bydgoszczy; Oddzial Kliniczny Onkologii, Bydgoszcz
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - RegioNAlny Osrodek Onkologiczny Pododdział Diagnostyki i Terapii Onkologicznej, Lodz
  - Regionalny Osrodek Onkologiczny; Oddzial Chorob Rozrostowych, Lodz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej; Opolskie Centrum Onkologii, Opole
  - Centrum Onkologii - Instytut, Klinika Nowotworow Tkanek Miekkich, Kosci i Czerniakow, Warsaw
- Sweden (2):
  - Blekingesjukhuset; Kirurgkliniken, Karlskrona
  - Karolinska University Hospital;Department of Oncology-Pathology, Stockholm
- United Kingdom (13):
  - Royal Sussex County Hospital, Brighton
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrookes Hospital; Dept of Oncology, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Cheltenham General Hospital; Gloucestershire Oncology Centre, Cheltenham
  - Dorset County Hospital NHS Foundation Trust;Research and Development/ Oncology, Dorchester
  - St James University Hospital, Leeds
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - St George's Hospital; Oncology, London
  - Imperial College Healthcare NHS Trust;Medical Oncology, London
  - The Clatterbridge Cancer Ctr For Oncolgy, Metropolitan Borough of Wirral
  - St Helens & Knowsley Trust, St Helens
  - New Cross Hospital; Deansley Centre, Wolverhampton